CLINICAL TRIAL: NCT01576068
Title: Efficiency of COPD Case Finding Program by Spirometry in High-risk Customers of Urban Community Pharmacies
Brief Title: Chronic Obstructive Pulmonary Disease Case Finding in Community-pharmacies by Spirometry
Acronym: FARMAEPOC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Col·legi de Farmacèutics de la Província de Barcelona (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Clinic of Barcelona (Other); Spanish Respiratory Society (Other); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008/3128/I
Record Dates: First submitted 2012-02-29; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pharmacy; Spirometry; Case finding
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Risk Customers (Other): Pharmacy customers with GOLD COPD Criteria of high-risk subjects.
  Interventions: Other: Spirometry

INTERVENTIONS:
Other: Spirometry — Spirometry done in high-risk customers of community-pharmacies to detect airflow limitation

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a prevalent disease. In the investigators country, underdiagnosis has been estimated in around 80% of subjects. Early detection is done mainly in primary care but due to actual situation new alternatives have been proposed to decrease underdiagnosis.

This present study promote by a multidisciplinary research team (respiratory medicine, primary care, nurse and pharmacist) raise the objective of evaluate the effect of a COPD case finding program guide by spirometry in community-pharmacies.

From the results of a pilot-study conducted in 13 community-pharmacies in Barcelona, in which the investigators showed the feasibility of spirometry in community-pharmacies for the early detection of COPD, the investigators have design a second phase to evaluate the effect of this strategy. 100 Barcelona's community-pharmacies during 6 months will select high risk customers and will conduct a spirometry in agreement with the design protocol. 3600 spirometries is the establish objective. Participants hospitals will train pharmacist in spirometry and also control spirometry quality daily by a telematic pathway. Spirometry results will be evaluate in terms of effect and costs. The investigators will also evaluate the impact of this program in the health system by numbers of subjects diagnosed and follow up in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years.
* Current or former smoker
* Chronic respiratory symptoms(cough, shortness of breath, expectoration)

Exclusion Criteria:

* Previous diagnosed chronic lung disease
* Use of inhalers

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-07 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
COPD Case Finding | During 15 months pharmacies will include subjects with possible COPD through spirometry.
  Proportion of high-risk customers with spirometry showing a FEV1/FVC under 0,7.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Castillo, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Col·legi Oficial de Farmacèutics de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Castillo D, Guayta R, Giner J, Burgos F, Capdevila C, Soriano JB, Barau M, Casan P; FARMAEPOC group. COPD case finding by spirometry in high-risk customers of urban community pharmacies: a pilot study. Respir Med. 2009 Jun;103(6):839-45. doi: 10.1016/j.rmed.2008.12.022. Epub 2009 Feb 5. PMID 19200706